CLINICAL TRIAL: NCT03622502
Title: The Effect of Dexmedetomidine on the Remifentanil Concentration for Preventing Cough During Emergence After Propofol Anesthesia
Brief Title: The Effect of Dexmedetomidine for Emergence Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AJIRB-MED-OBS-18-170
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Cough
Keywords: dexmedetomidine; remifentanil; extubation
MeSH Terms: conditions — Cough | interventions — Dexmedetomidine; Remifentanil; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine was infused before end of surgery and remifentanil was maintained at predetermined effect-site concentration during the emergence period
  Interventions: Drug: Dexmedetomidine; Drug: Remifentanil
- Remifentanil (Active Comparator): Normal saline was infused before end of surgery and remifentanil was maintained at predetermined effect-site concentration during the emergence period
  Interventions: Drug: Remifentanil; Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 0.5mcg/kg was infused over 10 min before end of the surgery
  Other Names: Prededex
  Arms: Dexmedetomidine
Drug: Remifentanil — Remifentanil was maintained at predetermined effect-site concentration during the periextubation period (initial concentration: 2.0 ng/ml)
  Other Names: Ultiva
Drug: Normal saline — Normal saline was infused over 10 min before end of the surgery
  Other Names: 0.9% NaCl
  Arms: Remifentanil

SUMMARY:
Dexmedetomidine or remifentanil are effective in attenuating cough during peri-extubation period after general anesthesia. The purpose of this study was to investigate the effect of dexmedetomidine on the remifentanil concentration for the cough suppression during anesthetic emergence.

DETAILED DESCRIPTION:
Administration of dexmedetomidine before end of surgery could reduce airway reflexes and hemodynamic changes during tracheal extubation. Compared with remifentanil alone, administration of dexmedetomidine in combination with remifentanil is effective in relieving cough and hemodynamic changes without inhibition of respiration. The purpose of this study was to investigate the effect of dexmedetomidine on the remifentanil concentration for the cough suppression during anesthetic emergence using the modified up-and-down method.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II undergoing endoscopic sinus surgery or septoplasty under general anesthesia

Exclusion Criteria:

* predicted difficult airway
* body mass index > 35 kg/m2,
* recent upper respiratory infection
* asthma
* current smoker
* patients using angiotensin converting enzyme-inhibitors
* uncontrolled hypertension

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Number of cough | from end of surgery to 5 min after tracheal extubation]
  Number of cough or a strong and sudden contraction of the abdomen during periextubation periextubation periods

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, Principal Investigator — Ajou University Hospital, Suwon, Gyeongki-do, Korea
Locations (1):
- Ajou University Hospital, Suwon, Gyeongki-do, South Korea

REFERENCES:
- [Derived] Kim HY, Kwak HJ, Lee D, Lee JH, Min SK, Kim JY. Comparison of remifentanil concentrations with and without dexmedetomidine for the prevention of emergence cough after nasal surgery: a randomized double-blinded trial. BMC Anesthesiol. 2021 May 4;21(1):136. doi: 10.1186/s12871-021-01358-x. PMID 33941098